CLINICAL TRIAL: NCT06326125
Title: Randomized Controlled Trial Examining the Effectiveness of Pharmacology and Non-pharmacology Approaches in Reducing Children's Pain and Fear During Painful Procedures
Brief Title: Pharmacology and Non-pharmacology Approaches in Reducing Children's Pain and Fear During Painful Procedures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Sherzad Khudeida Suleman, Principal Investigator, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SherzadSH
Record Dates: First submitted 2024-02-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Pain
Keywords: pain, anxiety, painful procedures
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- TICK-B (Experimental): active distraction technique as non-pharmacology in treating children's pain and fear during venipuncture procedure.
  Interventions: Behavioral: TICK-B
- TkTx-Cream (Experimental): as Pharmacological approach will be use in managing children's pain and fear during venipuncture procedure.
  Interventions: Drug: TKTX-Cream
- TICK-B and TkTx-C (Experimental): Pharmacological approache and non-Pharmacological will be use in managing children's pain and fear during venipuncture procedure.
  Interventions: Other: TICK-B and TKTX-C
- Control Group (No Intervention): No intervention will applied in this group

INTERVENTIONS:
Behavioral: TICK-B — TICK-B as art-based distraction
  Arms: TICK-B
Drug: TKTX-Cream — TKTX-Cream as local anesthesia cream
  Other Names: Local anesthesia
  Arms: TkTx-Cream
Other: TICK-B and TKTX-C — TICK-B and TkTx-C as combined intervention approche (pharmacology and non-pharmacology)
  Other Names: Combination approach
  Arms: TICK-B and TkTx-C

SUMMARY:
This study Will contribute in the knowledge of pediatric nurses during painful procedures such venipuncture

DETAILED DESCRIPTION:
Children frequently undergo unexpected and procedure-related pain while in hospital settings, leading to adverse emotional and psychological effects. The exposure to painful procedures, particularly venipuncture, commonly occurs in emergency units, upon admission, during hospital stays, or during follow-up visits. The mere act of inserting needles stands out as one of the most distressing medical procedures for children, resulting in frightening and upsetting experiences for both the children and their parents throughout the hospitalization period.

In the realm of pain management, interventions can generally be classified into pharmacological and non-pharmacological approaches. Within pharmacological interventions, local anesthetics play a key role in addressing needle-related pain. These anesthetics can permeate the cuticle and epidermal layers of intact skin, reaching the dermis where nerve endings are situated, thereby alleviating pain. Notably, a eutectic mixture of local anesthetics (EMLA) emulsion, composed of 25 mg lidocaine and 25 mg prilocaine per gram, has been explored in pediatric settings for managing venipuncture pain due to its effectiveness and minimally invasive nature.

On the non-pharmacological front, various strategies have been investigated for needle procedures in children, including distraction techniques, cognitive and behavioral therapy, hypnosis, and memory alteration. Among these interventions, distraction stands out as a straightforward method that can be promptly applied and requires minimal prior training. A systematic review has demonstrated the effectiveness of distraction in alleviating pain associated with needle-related procedures.

ELIGIBILITY:
Inclusion:

School-aged 6-12 years old. Children who require PIVC.

Exclusion:

1. Chronic diseases,
2. Physical impairment,
3. Disability contributes to difficult communication,
4. Children of unsatisfied parents,
5. Children with neurodevelopment delays,
6. Cognitive impairment, hearing impairment, or visual impairment,
7. Taking an analgesic within 6 hours, or those with a syncope history.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-04-10 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
severity of Pain | baseline, during, and immediately post-procedure.
  Severity of pain will be assessed using Wong-Baker FACES Pain Rating Scale, a validated self-reporting tool widely utilized in clinical settings. Participants will be instructed to rate their pain on a scale from 0 (indicating no pain) to 10 (representing the worst imaginable pain). The Wong-Baker FACES Pain Rating Scale will be administered promptly after the completion of the procedure.

SECONDARY OUTCOMES:
Fear | baseline, during, and immediately post-procedure.
  level of fear will be assessed using the Child Fear Scale (CFS), a validated instrument designed to measure the level of fear in pediatric populations. Participants will be asked to express their feelings of fear related to the procedure through the Child Fear Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sherzad Suleman, MsC, Principal Investigator — Uppsala University
Locations (1):
- Sherzad Khudeida Suleman, Duhok, Erbil Governorate, Iraq

REFERENCES:
- [Derived] Suleman SK, Yahya N, Nilsson S, Enskar K. Comparative efficacy of pharmacological and non-pharmacological interventions for mitigating pain and anxiety associated with venipuncture: a randomised controlled trial. BMJ Paediatr Open. 2024 Sep 9;8(1):e002881. doi: 10.1136/bmjpo-2024-002881. PMID 39251366